CLINICAL TRIAL: NCT06651541
Title: Phase 2 Parallel Clinical Study to Evaluate the Efficacy in Increasing Sexual Arousal, Safety and Tolerability of BZ371A in Gel Form Applied to Women With Sexual Arousal Disorder
Brief Title: Evaluation of the Efficacy in Increasing Sexual Arousal, Safety and Tolerability of BZ371A in Women With Sexual Arousal Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biozeus Biopharmaceutical S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BZ371CLI602
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Female Sexual Arousal Disorder; Female Sexual Dysfunction (FSD)
Keywords: sexual dysfunction; Topical application; female
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BZ371A group (0.5 ml) (Experimental): The medication will be administered at least twice a week (according to demand), followed by sexual encounters, for 8 weeks
  Interventions: Drug: BZ371A (0.5 ml); Drug: Placebo (0.5 ml)
- Placebo Group (0.5 ml) (Placebo Comparator): The medication will be administered at least twice a week (according to demand), followed by sexual encounters, for 8 weeks
  Interventions: Drug: BZ371A (0.5 ml); Drug: Placebo (0.5 ml)
- Placebo Group (1.0 ml) (Placebo Comparator): The medication will be administered at least twice a week (according to demand), followed by sexual encounters, for 8 weeks
  Interventions: Drug: Placebo (1.0 ml); Drug: BZ371A (1.0 ml)
- BZ371A group (1.0 ml) (Experimental): The medication will be administered at least twice a week (according to demand), followed by sexual encounters, for 8 weeks
  Interventions: Drug: Placebo (1.0 ml); Drug: BZ371A (1.0 ml)

INTERVENTIONS:
Drug: BZ371A (0.5 ml) — Formulation with the active ingredient
  Arms: BZ371A group (0.5 ml); Placebo Group (0.5 ml)
Drug: Placebo (0.5 ml) — Formulation without the active ingredient
  Arms: BZ371A group (0.5 ml); Placebo Group (0.5 ml)
Drug: Placebo (1.0 ml) — Formulation without the active ingredient
  Arms: BZ371A group (1.0 ml); Placebo Group (1.0 ml)
Drug: BZ371A (1.0 ml) — Formulation with the active ingredient
  Arms: BZ371A group (1.0 ml); Placebo Group (1.0 ml)

SUMMARY:
Evaluation of the efficacy in increasing sexual arousal, safety and tolerability of BZ371A in gel form applied to women with sexual arousal disorder

DETAILED DESCRIPTION:
Female Sexual Arousal Disorder (FSAD) is defined as the recurrent inability to attain or maintain sufficient genital arousal during sexual activity. Therefore, a healthy blood flow is central to the physiological processes related to sexual arousal, leading to genital lubrication, warmth, and clitoral protrusion.

The vasculature and blood flow in vaginal tissue can be compromised due to natural aging and various risk factors, including cigarette smoking, alcohol abuse, lack of exercise, high-fat diets, hypertension, hypercholesterolemia, and diabetes mellitus. All these risk factors and conditions are highly prevalent among women and can lead to FSAD. BZ371A offers a potential solution by increasing blood flow in genital tissue through its unique mechanism of action, thereby restoring vascular homeostasis and the physiological processes related to sexual arousal in women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 21 and 65 years;
* Premenopausal or postmenopausal women may be included;
* May or may not be using female sex hormones (estrogen with or without progesterone, or their derivatives);
* Women who have previously had sexual experiences with orgasm, desire, and arousal, for a minimum period of two years;
* FSD, defined according to DSM-IV diagnostic criteria, that is, the presence of a persistent or recurrent inability to achieve or maintain adequate physiological sexual arousal during sexual activity, meaning a reduction or absence of genital response (lubrication, clitoral swelling, or other genital responses such as genital pleasure sensations);
* FSD causes significant personal distress and/or interpersonal difficulty;
* FSFI questionnaire meeting criteria for female sexual dysfunction, i.e., <26.5;
* Stable relationship for more than 6 months, with a sexually active partner who is present (cannot be traveling, for example) during the treatment period;
* Ability to read and understand the Informed Consent Form (ICF) and to complete the questionnaires.

Exclusion Criteria:

* Women who do not agree to use a contraceptive method and who have the capacity to become pregnant during the study;
* Women who do not agree to attempt sexual activity at least twice a week while taking the study medication;
* Serious relationship problems, defined as a CSI-16 score below 51.5, of non-sexual origin, and which, in the investigator's opinion, may influence sexual activities;
* History of unresolved sexual trauma or abuse, that could interfere with participation or the results of the study;
* Diagnosis of vaginismus, genitopelvic pain/penetration disorder and/or sexual aversion disorder;
* Uncontrolled diabetes at screening visit (HbA1C > 10%);
* Prior spinal cord injury, with lower limb paralysis;
* History of abdominal or pelvic surgery that may have damaged pelvic nerves, including vulvectomy, colostomy, cytostomy, hysterectomy, or bladder suspension;
* Current testosterone use, or long-term testosterone use (such as chip) within the past 6 months;
* Patients with severe current depression, characterized by the use or need for the use of psychotropic medications, including bupropion, lithium, or neuroleptics (patients using antidepressant medications such as selective serotonin reuptake inhibitors may participate);
* Presence of genital lesions that impair analysis of local adverse effects on the genitalia;
* Presence of diseases that cause excessive vaginal discharge, such as recurrent urinary tract infection, vaginal infection and pelvic inflammatory disease.
* Abnormal Papanicolaou test within the past 3 years;
* History of gynecological cancer (history of uterine dysplasia can be included, provided it has been properly treated for at least 6 months);
* History of pelvic irradiation;
* Use of topical medications in the genital region that may interfere with PSI assessment as well as their absorption or drug interaction, including vaginal estrogens, lubricants, spermicides, creams or gels, vaginal douches;
* History of symptomatic hypotension, or diseases that increase the risk of symptomatic hypotension, such as patient with heart disease (including history of angina and/or heart failure) and nephropathies;
* Current use of nitrates, such as propatylnitrate (Sustrate®), isosorbide (Monocordil®, Cincordil®, Isordil®), nitroglycerin (Nitradisc®, Nitroderm TTS®, Nitronal®, Tridil®) and isosorbitol dinitrate (Isocord®)
* ECG findings that are clinically symptomatic, or that, in the Investigator's judgment, are considered significant and pose a risk to the research volunteer's participation;
* Findings on laboratory tests that, in the Investigator's judgment, are considered significant and offer risk to the research volunteer's participation or may hinder the study analyses;
* TSH outside the normal range for age and/or participants with hypothyroidism who started thyroid hormone replacement less than 3 months ago, even if TSH is within normal limits;
* BP outside safe limits: SBP below 90 mmHg or above 170 mmHg; or DBP below 50 mmHg or above 100 mmHg, except for situations such as "white coat" syndrome;
* Severe hypertension, considered to be the use of three or more antihypertensive drugs;
* Diseases that can cause clitoral priapism, such as sickle cell anemia, multiple myeloma or leukemia;
* History of clitoral priapism;
* Current relevant diarrhea, defined as duration over four weeks, association with abdominal pain or malabsorptive syndrome, or presence of mucus, pus, or blood in the stool;
* Pregnant or lactating;
* Current use of nitric oxide donors, guanylate cyclase stimulators (e.g. Riociguat), or 5- phosphodiesterase inhibitors (Sildenafil, Tadalafil, etc.);
* Any disease or condition or physical finding that the Investigator considers significant and that increases the risk of the research participant's participation or may interfere with the results, including serious debilitating diseases, presence of cancer, serious mental illness, persistent abuse of medication;
* Partners with significant erectile dysfunction, defined as the inability to maintain an erection to provide satisfactory sexual intercourse in most sexual encounters;
* Having participated in the BZ371CLI601 study;
* Known hypersensitivity to BZ371A or any of the components of the formulation;
* Significant tobacco or alcohol abuse that, in the investigator's opinion, may impair the participant's sexual function (light or moderate use of tobacco or alcohol is permitted);
* Less than 3 valid sexual encounters, defined as a "yes" answer to question 7 of the FSEP, or use of less than 3 doses of PSI in the run-in period.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — heterosexual
Enrollment: 174 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy in increasing arousal | Baseline, 4 weeks and 8 weeks
  Evaluation of the efficacy of BZ371A in increasing arousal using Female Sexual Encounter Profile (FSEP) questionnaire. The study will evaluate number of "yes" answers to question 3 in the Female Sexual Encounter Profile (FSEP) questionnaire, divided by the number of valid attempts (question 7 of the FSEP).
  The study will evaluate the increase in the FSEP score based on the baseline FSEP value, obtained before using the BZ371A. Thus, the higher the number of yes answers, the better the efficacy of the drug.

SECONDARY OUTCOMES:
Efficacy in increasing desire, lubrification, orgasm and arousal | Baseline, 4 weeks and 8 weeks
  Evaluation of the success rate for desire, lubrification, orgasm and for arousal using Female Sexual Encounter Profile (FSEP). The number of successes for desire will be assessed using FSEP Question 2 / FSEP Question 7, for lubrication FSEP Question 4 / FSEP Question 7, for orgasm FSEP Question 5 / FSEP Question 7 and for the degree of arousal FSEP Question 6 / FSEP Question 7. For each question, the number of "yes" answers will be counted as success. Therefore, for each "no" answer the value will be 0 and for each "yes" answer the value will be 1.
Evaluation of the quality of female sexual encounters | Baseline, 4 weeks and 8 weeks
  Evaluation based on the total score of the Female Sexual Encounter Profile (FSEP) questionnaire. The score ranges from 0 to 9. Therefore, the higher the score, the better the participant's sexual encounter.
Female Sexual Function Index (FSFI) | Baseline, 4 weeks and 8 weeks
  Evaluation of the score for each domain (Desire, Arousal, Lubrication, Orgasm, Satisfaction, Pain) using the Female Sexual Function Index (FSFI) questionnaire. The score ranges from 2 to 36. Thus, the higher the score, the better the participant's sexual satisfaction.
Assessment of treatment satisfaction | Baseline, 4 weeks and 8 weeks
  Response rate to the Global Assessment Question (GAQ), by the number of "yes" answers to the question about arousal and sexual pleasure.
Adverse effects report | Baseline, 4 weeks, 8 weeks and 10 weeks after baseline
  Adverse effects evaluation of compound use and application
Physical examination of the genitalia | Up to 60 days before baseline, 30 days before baseline, baseline, 4 weeks, 8 weeks and approximately 11 weeks
  Number of participants with abnormal physical exam findings in the applied region.
Change in systemic blood pressure | From up to 60 days before Baseline, 30 days before Baseline, Baseline, 4 weeks, 8 weeks and, approximately, 10 weeks
  Change in Diastolic Blood Pressure and Systolic Blood Pressure
Change in Heart Rate (HR) | From up to 60 days before Baseline, 30 days before Baseline, Baseline, 4 weeks, 8 weeks and, approximately, 11 weeks
  Change in Heart Rate
Basal chest electrocardiogram (ECG) | From up to 60 days before baseline, baseline and 8 weeks after baseline
  Number of participants with abnormal electrocardiogram (ECG) findings.
Blood evaluation | From up to 60 days before Baseline, baseline and 8 weeks after baseline
  Number of participants with abnormal laboratory test results
Urine evaluation | From up to 30 days before baseline, baseline and 8 weeks after baseline
  Number of participants with abnormal laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Fabiene Vale, MD PhD, Principal Investigator — Hospital das Clínicas - UFMG
Locations (1):
- Ambulatório Jenny Farias do Hospital das Clínicas da UFMG, Belo Horizonte, Brazil

IPD SHARING:
Plan to Share IPD: No